CLINICAL TRIAL: NCT01123434
Title: A Non-interventional Study of Immediate Postoperative Adjuvant Hormonal Treatment in High Risk Localised or Locally Advanced Chinese Prostate Cancer Patients.
Brief Title: Immediate Postoperative Adjuvant Hormonal Treatment in High Risk Localised or Locally Advanced Prostate Cancer Patients.
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OCN-DUM-2009/2
Record Dates: First submitted 2010-05-10; First posted 2010-05-14 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: 2 Years PSA Recurrence Rate
Keywords: prostate cancer; adjuvant; hormonal
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Localised with one of any high recurrence risk factors, or locally advanced Chinese prostate cancer patients confirmed histologically through radical prostatectomy either with laparoscopy or laparotomy within 1 month after surgery. Before the patient recruitment, the investigator has decided to prescribe immediate postoperative adjuvant hormonal treatment to the patient according to the Chinese routine practice.

SUMMARY:
The primary objective is to assess the efficacy of immediate postoperative adjuvant hormonal treatment according to 2 year PSA recurrence rate in high risk localised or locally advanced Chinese prostate cancer patients.The secondary objective is to assess the quality of life（QoL）of the high risk localised or locally advanced Chinese prostate cancer patients with immediate postoperative adjuvant hormonal treatment and get the information of immediate postoperative adjuvant hormonal treatment (including the regimen, dosage and duration).

ELIGIBILITY:
Inclusion Criteria:

* Localised with one of any high recurrence risk factors(Gleason score≥8 or preoperative serum PSA≥20ng/ml), or locally advanced(T≥pT3、N0M0 and any T、N（+）M0 ) Chinese prostate cancer patients confirmed histologically through radical prostatectomy either with laparoscopy or laparotomy within 1 month after surgery. Before the patient recruitment, the investigator has decided to prescribe immediate postoperative adjuvant hormonal treatment to the patient according to the Chinese routine practice.
* Provision of written informed consent prior to any study specific procedures.

Exclusion Criteria:

* Patients must not enter the study if any of the following exclusion criteria are fulfilled
* Have used neoadjuvant hormonal treatment prior to the surgery.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients form urology surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of immediate postoperative adjuvant hormonal treatment according to 2 year PSA recurrence rate in high risk localised or locally advanced Chinese prostate cancer patients. | Up to 2 years

SECONDARY OUTCOMES:
To assess the quality of life（QoL）of the high risk localised or locally advanced Chinese prostate cancer patients with immediate postoperative adjuvant hormonal treatment. | Up to 2 years
Get the information of immediate postoperative adjuvant hormonal treatment (including the regimen, dosage and duration). | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Karen Atkin, Study Director — AstraZeneca; Yanjing Zhang, Study Chair — AstraZeneca; Prof. Na, Principal Investigator — Peking University Shougang Hospital; Prof. Ye, Principal Investigator — Tong Ji Hospital of Tongji Medical College of Huazhong University of Science and Technology
Locations (10):
- China (10):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Wuhan, Hubei
  - Research Site, Nanjing, Jiangsu
  - Research Site, Shenyang, Liaoning
  - Research Site, Xi’an, Shanxi
  - Research Site, Chengdu, Sichuan
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Shanghai
  - Research Site, Tianjin